CLINICAL TRIAL: NCT01458132
Title: WEUSKOP5522: Observational Drug Exposure Registry for Long-Term Follow-Up of Subjects Exposed to GSK2248761
Brief Title: Drug Exposure Registry for GSK2248761, an Investigational NNRTI
Status: Completed | Type: Observational
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 115682; WEUSKOP5522 (Other: GSK); EPI40670 (Other: GSK)
Record Dates: First submitted 2011-09-01; First posted 2011-10-24 (Estimated); Results first posted 2019-09-11 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-07

CONDITIONS: HIV Infections
Keywords: subject follow-up; HIV infection; registry; seizures; GSK2248761
MeSH Terms: conditions — HIV Infections; Seizures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects who experienced seizure: Subjects who were previously randomized in the Phase 2b studies SGN113399 or SGN113404 and experienced seizure
- Subjects who did not experience seizure: Subjects who were previously randomized in the Phase 2b studies SGN113399 or SGN113404 and did not experience seizure

SUMMARY:
The World Health Organization has estimated that as many as 10% of the population worldwide may at some point experience at least one seizure. The percentage with active epilepsy is from 0.4% to 1%. From 40% to 65% of patients with HIV infection have been estimated to have some neurological involvement; the percentage reaches as high as 70% to 80% when post-mortem assessments are included. Estimates of the percentage of HIV-infected patients with seizure occurrence have varied widely, with one review finding a range from 2% to 20%. The highest percentage in this range was reported at a center that exclusively treated patients with neurological involvement, in India where HIV clade C subtype is predominant. Query of another neurology department's database determined that of the HIV-infected patients treated at the center, all of whom were referred for neurological symptoms, 6.1% experienced seizures. Underlying neurologic diseases in these patients included HIV-associated encephalopathy, progressive multifocal leukoencephalopathy, and toxoplasmosis. In a Spanish population, 3% of HIV-infected patients over a one-year study period were found to have new-onset seizures, which were attributed to drug toxicity in 47%, intracranial lesions in 35%, and metabolic derangements in 12%.

Drug-discontinuation studies, magnetic resonance imaging studies, and animal studies have produced recent evidence that some antiretroviral therapies may have neurotoxic effects, warranting further research. Individuals who are treated with highly active antiretroviral therapy are at risk for immune reconstitution inflammatory syndrome (IRIS), in which immune recovery triggers clinical deterioration as the newly invigorated immune system reacts to pathogens that either represent ongoing opportunistic infection or were previously successfully controlled. In a population initiating combination antiretroviral therapy between 1999 and 2007, 0.9% developed neurological manifestations of IRIS. Seizures may occur as part of a neurological IRIS syndrome, such as encephalitis and toxoplasmosis.

Two randomized, Phase 2b dose-finding studies were conducted in HIV-1 infected adults to compare GSK2248761 100 mg and 200 mg given once daily as part of an antiretroviral treatment regimen. One of the studies (SGN113399) was in subjects with prior exposure to antiretroviral therapy where GSK2248761 100 mg and 200 mg once daily were compared to determine the best dose in this population. A contemporary control arm receiving etravirine 200 mg twice daily was also included, and all arms included a twice-daily background therapy consisting of darunavir/ritonavir 600 mg/100 mg plus raltegravir 400 mg. The other study (SGN113404) was in treatment-naïve subjects, comparing GSK2248761 100 mg and 200 mg once daily to determine the best dose in this population. A contemporary control arm receiving efavirenz 600 mg once daily was also included, and all arms were given background therapy selected by investigators from either once-daily abacavir/lamivudine 600 mg/300 mg or tenofovir/emtricitabine 300 mg/200 mg. Of a planned total population in both studies of 300 subjects, 35 were enrolled before the studies were terminated because of the occurrence of seizures in five subjects. All of the subjects who experienced seizures were enrolled into SGN113399, four randomized to receive 200 mg GSK2248761 and one randomized to receive 100 mg GSK2248761. There were no seizures in the subjects receiving GSK2248761 in study SGN113404. At the time of study termination, subjects had been enrolled and received GSK2248761 at 19 sites in four countries: France, Romania, United States, and Germany. Although potential contributory conditions have been identified in some cases, definitive causative factors for the seizure occurrence have not been established.

The purpose of this study is to follow subjects who previously received GSK2248761 while enrolled in the Phase 2b studies, which were halted due to unexpected seizures. The study will collect data on all subjects and will be used to monitor for additional seizures as well as collect additional clinical data on all subjects.

DETAILED DESCRIPTION:
The objective of the study is to collect and monitor data on all subjects who previously received GSK2248761 while enrolled in the Phase 2b studies SGN113399 or SGN113404 evaluating GSK2248761. There will be no formal hypotheses tested, and the data collected will be utilized to build individual subject narratives for each subject.

All subjects who were previously randomized in the Phase 2b studies SGN113399 or SGN113404 and received GSK2248761, will be targeted for enrollment in the study. Study SGN11339 had 20 subjects randomized to receive GSK2248761 and was conducted at 12 sites in the United States and one site in Romania. Study SGN113404 was conducted at three sites in France and three sites in Germany, with 15 subjects randomized to receive GSK2248761. Therefore, the study population for the current study will consist of 35 subjects originating from sites located in the United States, Romania, France, and Germany.

All subjects enrolled in this study previously received GSK2248761 in one of the Phase 2b clinical trials SGN113399 or SGN113404 of GSK2248761 for the treatment of HIV. This study will collect clinical and safety data on all subjects. Data from these subjects' medical charts will be collected from the point of termination of the Phase 2b clinical trials. Any subject who experienced any seizure during the Phase 2b clinical trial will be followed for two years. Subjects who experienced no seizure during the Phase 2b clinical trial will be followed for one year. In the event that a subject who did not previously have a seizure experiences a seizure during the study period, the subject will be moved to the "seizure subject group" that is being followed for two years. Data collection will occur on a quarterly basis for all subjects.

No formal analyses will be performed. All data collected for each subject will be incorporated into a narrative of the subject's medical events during the follow-up period. The narrative will recreate the clinical course and evolution of disease history for the subjects and allow assessment for evidence of residual or new adverse events potentially related to their exposure to GSK2248761. Listings of AEs will be generated for each subject. Data on AEs collected quarterly will be combined with the subject's demographic and medical history details in the listing reports. The listings will be delivered to GSK every six months in coordination with the safety advisory committee meetings.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who were previously randomized in the Phase 2b studies SGN113399 or SGN113404 and received GSK2248761

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All subjects who were previously randomized in the Phase 2b studies SGN113399 or SGN113404 and received GSK2248761 will be targeted for enrollment in the study. Study SGN11339 had 20 subjects randomized to receive GSK2248761 and was conducted at 12 sites in the United States and one site in Romania. Study SGN113404 was conducted at three sites in France and three sites in Germany, with 15 subjects randomized to receive GSK2248761. Therefore, the study population for the current study will consist of 35 subjects originating from sites located in the United States, Romania, France, and Germany.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2011-07-29 (Actual); Primary Completion 2013-04-30 (Actual); Study Completion 2013-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 06 September 2011 to 25 February 2013, at 19 sites in 4 countries, France, Romania, United States, and Germany.
Pre-assignment Details: Of the 35 Fosdevirine -exposed participants, 19 consented to enroll in the registry, including 4 of the 5 seizure participants and 15 from the non-seizure group.
Groups:
- Participants Without Seizure: Participants who were previously randomized in the Phase 2b studies SGN113399 or SGN113404 (randomized to Fosdevirine) and did not experience seizure during the follow-up period, after exposure to Fosdevirine, at 100 or 200 milligram (mg), for atleast four weeks in the Phase 2b trials.
- Participants With Seizure: Participants who were previously randomized in the Phase 2b studies SGN113399 or SGN113404 and experienced seizure during the follow-up period , after exposure to fosdevirine, at 100 or 200 mg, for atleast four weeks in the Phase 2b trials.
Period: Overall Study
Arm/Group | Participants Without Seizure | Participants With Seizure
Started | 15 | 4
Completed | 0 | 1
Not Completed | 15 | 3
Not completed — Other | 15 | 3

BASELINE CHARACTERISTICS:
Population: All Subject Population: all participants who consented to participate in the registry study.
Groups:
- Participants Without Seizure: Participants who were previously randomized in the Phase 2b studies SGN113399 or SGN113404 (randomized to Fosdevirine ) and did not experience seizure during the follow-up period, after exposure to Fosdevirine, at 100 or 200 mg, for atleast four weeks in the Phase 2b trials.
- Total: Total of all reporting groups
Arm/Group | Participants Without Seizure | Participants With Seizure | Total
Number analyzed (Participants) | 15 | 4 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 4 | 19
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 12 | 3 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Occurrence of Seizure
Description: In the registry study from start to the end of follow-up, the number of participants who experienced seizure were reported. This was done to evaluate to test the time-efficiency and cost-efficiency for a long term, non-interventional study.
Time Frame: Up to 17 months
Population: All Subject Population, defined as all participants, who consented to participate in the registry study.
Measure: Count of Participants; unit: Participants
Groups:
- Participants Without Seizure: Participants who were previously randomized in the Phase 2b studies SGN113399 or SGN113404 (randomized to Fosdevirine) and did not experience seizure during the follow-up period, after exposure to Fosdevirine, at 100 or 200 mg, for atleast four weeks in the Phase 2b trials.
- Participants With Seizure: Participants who were previously randomized in the Phase 2b studies SGN113399 or SGN113404 (randomized to Fosdevirine) and experienced seizure during the follow-up period, after exposure to fosdevirine, at 100 or 200 mg, for atleast four weeks in the Phase 2b trials.
Arm/Group | Participants Without Seizure | Participants With Seizure
Number analyzed (Participants) | 15 | 4
Participants | 0 | 1

2. Secondary Outcome: Number of Participants With Serious Adverse Event (SAE) and Adverse Event (AE)
Description: An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product. For marketed medicinal products, this also includes failure to produce expected benefits (i.e. lack of efficacy), abuse or misuse. SAE was any experience that: resulted in death, was life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect or was medically significant.
Time Frame: Upto 17 months
Population: All Subject Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Without Seizure | Participants With Seizure
Number analyzed (Participants) | 15 | 4
Participants
  Any AE | 15 | 4
  Any SAE | 1 | 0

ADVERSE EVENTS:
Time Frame: Up to 17 months
Description: All Subject Population was used
Arm/Group | Participants Without Seizure | Participants With Seizure
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/15 | 0/4
Other Adverse Events (participants affected / at risk) | 15/15 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants Without Seizure (N=15) | Participants With Seizure (N=4)
Staphylococcal infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Participants Without Seizure (N=15) | Participants With Seizure (N=4)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Eye abscess (Infections and infestations) | 1 | 0
Gastroenteritis salmonella (Infections and infestations) | 1 | 0
Hip arthroplasty (Surgical and medical procedures) | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0
Rhinitis allergic (Immune system disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Tobacco withdrawal symptom (Psychiatric disorders) | 1 | 0
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Vaginal infection (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.